CLINICAL TRIAL: NCT05686785
Title: Agreement and Reliability of Transient Elastography in Patients With Chronic Viral Hepatitis - a Cross-sectional Test-retest Study
Brief Title: Agreement and Reliability of Transient Elastography
Acronym: HEPSCAN
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: CIV-22-08-040567
Record Dates: First submitted 2022-12-07; First posted 2023-01-17 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Chronic Viral Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Chronic viral hepatitis
  Interventions: Diagnostic Test: Transient elastography

INTERVENTIONS:
Diagnostic Test: Transient elastography — Transient elastography measures liver stiffness in kPa
  Other Names: Fibroscan

SUMMARY:
The aim of this study is to assess agreement, smallest detectable change, and reliability of repeated measurements of liver stiffness of transient elastography in patients with chronic viral hepatitis, and to explore factors associated with disagreement.

DETAILED DESCRIPTION:
Previous studies have reported excellent test-retest reliability for transient elastography (TE) in viral hepatitis. Reliability refers the ability of an instrument to discriminate between study subjects and may be excellent even if considerable measurement-error exists, if the population is heterogenous. Agreement, in contrast, refers to differences of measurements on the original scale (kPa for TE). Whether agreement is acceptable is situation-dependent and can be related to the smallest detectable change (SDC).

Agreement metrics or SDC have not been addressed in previous studies for chronic viral hepatitis. The aim of this study is to assess agreement, SDC, and reliability of repeated measurements of liver stiffness of TE in patients with chronic viral hepatitis, and to explore factors associated with disagreement.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the departments of infectious diseases in Malmö, Lund and Helsingborg with chronic viral hepatitis.
* Adult patients
* Signed informed consent to participate in the study.

Exclusion Criteria:

* suspected or confirmed pregnancy.
* patients unable to speak Swedish
* inability to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic viral hepatitis, i.e. chronic hepatitis B (with or without chronic hepatitis D), of chronic hepatitis C.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Disagreement defined as a difference in TE results between operators in KPa of ≥ 33%, as well as the smallest detectable change, SDC95. | Assessed at a 30 min visit to the outpatient clinic
  Disagreement, expressed as 1) the proportion of participants with inter-rater differences at or above our prespecified threshold (33%) and 2) the smallest detectable change, representing the difference needed to state with 95% certainty that a change had occurred in the underlying fibrosis (SDC95).

SECONDARY OUTCOMES:
Reliability, estimated using the intra-class correlation | Assessed at a 30 min visit to the outpatient clinic
  Reliability, for continuous stiffness measurements as well as for different fibrosis stage categories.
Patient and exam characteristics associated with inter-rater differences above our prespecefied threshold. | Assessed at a 30 min visit to the outpatient clinic
  As an exploratory outcome, patient and exam characteristics associated with inter-rater differences above our prespecified threshold of ≥ 33% in liver stiffness will be evaluated. These characteristics include patients age, hepatitis b staging, BMI, biomarkers including Alanine transaminase, probe type, (medium or XL-probe) viral load, alkaline phosphatase, bilirubin, albumin, prothrombin time/international normalized ratio, time since food (hours), time since alcohol (hours), previous liver biopsy (years)

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Ljungquist, MD, PhD., Principal Investigator — Division of Infection Medicine, Department of Clinical Sciences, Lund University, Lund.
Locations (1):
- Oskar Ljungquist, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided